CLINICAL TRIAL: NCT04842721
Title: Effect of Prolonged Mouth Rinse With Hypertonic Saturated Saline Solution on the Naso-Pharyngeal Viral Load of Covid-19 Virus in Vivo.
Brief Title: Effect of Hypertonic Saturated Saline Mouth Rinse on Covid-19 Virus in Vivo.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Not yet meeting Health Canada's requirements for Clinical Trials
Sponsor: Rafik Batroussy (Other)
Responsible Party: Sponsor-Investigator, Rafik Batroussy, Principal Investigator, Batroussy, Rafik
Organization: Batroussy, Rafik (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2021-04-11; First posted 2021-04-13 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Covid19
Keywords: Rinse; Mouth Rinse; Mouthwash; Mouth Wash
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: A randomized blinded controlled study, whereas a number of patients (at least 20) with clinically-confirmed Covid-19 infection within 7 days prior to the start of the study, are equally divided into 2 groups, Active and Control groups, using Active and Control Mouth rinses respectively. The Active Rinse is a 25 ml of Hypertonic Saturated Saline solution made by mixing 10 grams of Sodium Chloride (Table Salt) in 25 ml of Tap water with some salt crystals deposited. The Control Rinse is a 25 ml of Plain Tap Water. Each Patient of both groups will be asked to keep the solution still in his/her mouth, close to the back of the mouth, for 30 minutes without gargling and without swallowing. After 30 minutes the solution will be spit out and mouth will be rinsed with plain water several times. The process will be done twice a day for 2 days. Patients of both groups will be tested once for Covid-19 7 days after the last treatment.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertonic Saturated Saline Mouth Rinse Active Arm (Active Comparator): The Active Rinse is a 25 ml of Hypertonic Saturated Saline solution made by mixing 10 grams of Sodium Chloride (Table Salt) in 25 ml of Tap water with some salt crystals deposited.
  Interventions: Drug: Hypertonic Saturated Saline Mouth Rinse Active Arm
- Plain Water Control Arm (Placebo Comparator): The Control Rinse is a 25 ml of Plain Tap Water.
  Interventions: Other: Placebo Plain Water Mouth Rinse Arm

INTERVENTIONS:
Drug: Hypertonic Saturated Saline Mouth Rinse Active Arm — Each Patient of this groups will be asked to keep the solution still in his/her mouth, close to the back of the mouth, for 30 minutes without gargling and without swallowing. After 30 minutes the solution will be spit out and mouth will be rinsed with plain water several times. The process will be done twice a day for 2 days.
  Arms: Hypertonic Saturated Saline Mouth Rinse Active Arm
Other: Placebo Plain Water Mouth Rinse Arm — Each Patient of this groups will be asked to keep the water still in his/her mouth, close to the back of the mouth, for 30 minutes without gargling and without swallowing. After 30 minutes the water will be spit out. The process will be done twice a day for 2 days.
  Arms: Plain Water Control Arm

SUMMARY:
Sars-Cov2 virus is transmitted through the respiratory route and by direct contact with contaminated surfaces and subsequent contact with nasal, oral or ocular mucosa. Many studies have found that the oral cavity and specifically the saliva may be a high-risk route for SARS-CoV-2 infection. Thus, strategies reducing salivary viral load could contribute to reduce the risk of transmission. Furthermore, studies have shown that SARS-CoV persists for two days in oral mucous membranes before its diffusion to the lower respiratory tract. This offers an interesting preventive and therapeutic window of opportunity for the control of this disease. In addition, Naso-pharyngeal viral load was linked with lung disease severity in a study of 12 patients with pneumonia.**. Some current studies around the world, as listed on ClinicalTrials.gov, are testing the effect of some common mouth rinses/gargles on the Covid-19 viral load, including Chlorhexidine gluconate, Hydrogen peroxide Povidone Iodine, Saline (1.102% w/v, slightly hypertonic) and Alcohol.

This study aims to test whether Prolonged Hypertonic Saline Mouth Rinse would reduce/eliminate*** the viral load in the Oro- Naso-Pharyngeal cavity, and could therefore be used as a strategy to reduce transmission risk in clinical and social settings.

The investigator hypothesizes that COVID-19-positive participants who use Hypertonic Saline Prolonged Rinse treatment will have an reduction/elimination of their Covid viral load, will develop a negative Covid test 7 days after intervention completion and will improve their clinical symptoms, potentially reducing lung disease severity.

DETAILED DESCRIPTION:
The aim of this study is to determine if prolonged rinsing (30 minutes) of mouth without gargling using a Hypertonic Saturated Sodium Chloride solution would reduce/eliminate the Upper Respiratory viral load in Covid-19 infected patients compared to a placebo (Plain Water Rinse). Patients who have been tested positive for COVID-19 using Nucleic Acid Test via Nose or Throat Swabs within 7 days prior to the start of the trial will be instructed to use either of the two treatment arms (Active or Placebo) for 30 minutes twice daily for two days and retested for Covid 7 days after the last treatment

A randomized blinded controlled study, whereas a number of patients (at least 20) with clinically-confirmed Covid-19 infection within 7 days prior to the start of the study, are equally divided into 2 groups, Active and Control groups, using Active and Control Mouth rinses respectively. The Active Rinse is a 25 ml of Hypertonic Saturated Saline solution made by mixing 10 grams of Sodium Chloride (Table Salt) in 25 ml of Tap water with some salt crystals deposited. The Control Rinse is a 25 ml of Plain Tap Water. Each Patient of both groups will be asked to keep the solution still in his/her mouth, close to the back of the mouth, for 30 minutes without gargling and without swallowing. After 30 minutes the solution will be spit out and mouth will be rinsed with plain water several times. The process will be done twice a day for 2 days. Patients of both groups will be tested once for Covid-19 7 days after the last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Tested positive for Covid in the past 7 days
* Have the ability to perform mouth rinse twice daily for 2 days and to undergo Covid testing by Oro or Naso-Pharyngeal swabs.
* No need for a ventilator for oxygenation support
* Can understand and read English
* Lives in Alberta Canada

Exclusion Criteria:

* Requiring mechanical ventilation
* Unable to perform mouth rinses twice times daily for 2 days
* Patients that are tested negative for COVID-19
* Patients who have been eating or drinking within an hour before or after each session
* Use of an antiseptic mouthwash within 7 days prior or after the study
* Patient who are intubated or too sick to give consent for the study.
* Not able to speak in English or lacking the decision-making capacity to consent for study.
* Inability to comply with protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Negative Covid PCR test results | 7 days
  The number of Negative PCR tests post intervention will be compared between both the Active group and the Control group. The Hypertonic Saturated Mouth Rinse intervention will be considered effective in reducing/eliminating Covid presence in the Oro-Nasopharyngeal area if the PCR Covid tests performed 7 days post termination of the study have more statistically-significant negative results in the Active group than in the Control group..

SECONDARY OUTCOMES:
Number of Participants with Change in Clinical Symptoms | 7 days
  A change in Covid Clinical symptoms (like fever, shortness of breath, dry cough, reduced lung functions, ..) in both the Active and Control groups will be monitored and statistically analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Rafik Batroussy, BSc.Pharm., Principal Investigator — Independent
Locations (1):
- Rafik Batroussy, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Antiviral Activity of Reagents in Mouth Rinses against SARS-CoV-2 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7582358/
- See also: Viral load under detectable levels can result in a False Negative PCR Covid test — https://www.cnn.com/2020/11/03/health/covid-test-negative-contagious-wellness/index.html